CLINICAL TRIAL: NCT00141882
Title: Memantine in Patients With Chronic Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192944-004
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: memantine

SUMMARY:
Randomized double-masked clinical trial of memantine in patients with glaucoma

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma damage on examination of visual field and optic disc
* Good visual acuity (with glasses if needed)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1119 (Actual)
Dates: Start 1999-03; Primary Completion 2006-01 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Progression of glaucoma